CLINICAL TRIAL: NCT01353716
Title: A Phase I, Open-Label, Parallel-Group Study to Evaluate the Pharmacokinetics and Safety of Dolutegravir in Subjects With Renal Impairment and Healthy Matched Control Subjects (ING113125)
Brief Title: Dolutegravir Renal Impairment Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 113125
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Healthy subjects matched to the renal impaired subjects by gender, age and body mass index to the renal impaired subjects. There will be a screening visit within 30 days of dose, a single dose of study drug and a follow-up visit 7-10 days after the dose of study drug.
  Interventions: Drug: Dolutegravir 50 mg
- Cohort 2 (Experimental): Subjects with severe renal impairment. There will be a screening visit within 30 days of dose, a single dose of study drug and a follow-up visit 7-10 days after the dose of study drug.
  Interventions: Drug: Dolutegravir 50 mg

INTERVENTIONS:
Drug: Dolutegravir 50 mg — Dolutegravir is an experimental drug in the integrase inhibitor class of HIV medications. There will be a one single dose of 50 mg.
  Other Names: GSK1349572

SUMMARY:
Dolutegravir (DTG, GSK1349572) is an integrase inhibitor being developed for the treatment of human immunodeficiency virus (HIV)-1 infection by GlaxoSmithKline (GSK) on behalf of Shionogi-ViiV Healthcare LLC. DTG is metabolized primarily by uridine diphosphate glucuronyltransferase (UGT)1A1, with a minor role of cytochrome P450 (CYP)3A, and with renal elimination of unchanged drug being extremely low (< 1% of the dose). Fifty-three percent of the total oral dose is excreted unchanged in the feces but it is unknown if all or part of this is due to unabsorbed drug or some percentage of biliary excretion of the glucuronide conjugate which can be further degraded to form the parent compound in the gut lumen. The current Food and Drug Administration (FDA) draft guidance for renal impairment studies states that a pharmacokinetic (PK) study in patients with renal impairment should be conducted even for those drugs primarily metabolized or secreted in bile, because renal impairment can inhibit some pathways of hepatic and gut drug metabolism and transport.

This study is planned as an open label, single-dose, pharmacokinetic study to evaluate plasma DTG pharmacokinetics following oral administration to subjects with severe renal impairment (creatinine clearance < 30 ml/min) and matched healthy controls. Results from this study are expected to enable the development of appropriate dosing recommendations in patients with renal impairment.

DETAILED DESCRIPTION:
ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between the age of 18 and 70 years is eligible to enter and participate in this study if he/she is: A healthy subject with a creatinine clearance >90 mL/min who are free from clinically significant illness or disease OR A renally impaired subject with a creatinine clearance of < 30 mL/min and are considered clinically stable in the opinion of the principal investigator.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol <40 pg/ml (<147 pmol/L) is confirmatory] OR Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit.
* Body weight greater than or equal to 50 kg for men and women and BMI within the range 19- 38 kg/m2 for renally impaired subjects; healthy matched control subjects will be matched to BMI +/- 25% and must also remain in the BMI range of 19- 38 kg/m2.
* Provide a signed and dated written informed consent prior to study participation.

Exclusion Criteria:

A healthy subject will not be eligible for inclusion in this study if any of the following criteria apply:

* A positive Hepatitis B surface antigen or positive Hepatitis C antibody result at screening.
* A positive test for HIV antibody at screening.
* The subject has a positive pre-study drug screen. Drugs that will be screened for include amphetamines, barbiturates, cocaine, and PCP.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to dose administration in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the dose of study medication.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy and inflammatory bowel disease should be excluded. Subjects with a history of peptic ulceration or pancreatitis within the preceding 6 months of screening should be excluded. Subjects with previous gastrointestinal (GI) surgery (except appendectomy more than three months prior to study) should be excluded.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* ALT >1.5xULN; alkaline phosphatase or bilirubin ≥ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* The subject's systolic blood pressure is outside the range of 90-145mmHg, or diastolic blood pressure is outside the range of 45-95mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* Screening ECG parameters outside of protocol limits

A subject with severe renal impairment will not be eligible for inclusion in this study if any of the following criteria apply:

* Evidence of recent infection with Hepatitis B within preceding 6 months. Subjects with chronic Hepatitis B (duration>6 months) are eligible for enrolment.
* A positive test for HIV antibody at screening.
* Subjects receiving hemodialysis, peritoneal dialysis, or any other renal replacement therapy or other medical procedure that serves as a surrogate for renal function.
* The subject has a positive pre-study drug screen. Drugs that will be screened for include amphetamines, barbiturates, cocaine, and PCP.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Subjects with a pre-existing condition (except renal impairment) interfering with normal gastrointestinal anatomy or motility that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy and inflammatory bowel disease should be excluded. Subjects with a history of peptic ulceration or pancreatitis within the preceding 6 months of screening should be excluded. Subjects with previous gastrointestinal (GI) surgery (except appendectomy more than three months prior to study) should be excluded.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* ALT >1.5xULN; alkaline phosphatase or bilirubin ≥ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.
* The subject's systolic blood pressure is outside the range of 90-160mmHg, or diastolic blood pressure is outside the range of 45-95mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* Screening ECG parameters outside of protocol limits
* Subjects using any concurrent prohibited medication.
* Subjects with a change in dose regimen of medically required medication within the 2 weeks prior to dosing.
* Subjects with fluctuating or rapidly deteriorating renal function. Assessment of the stability of the subject's renal function will be determined by the investigator.
* Subjects whose serum potassium levels are more than or equal to 6 mEq/L.
* Subjects whose serum sodium levels are less than or equal to 125 mEq/L.
* Subjects with signs of active infection.
* Subjects with any other medical condition which, in the judgement of the investigator and medical monitor, could jeopardize the integrity of the data derived from that subject or the safety of the subject.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Plasma PK parameters of DTG: Lag time before observation of drug concentrations in sampled matrix (tlag) | 72 hours
Plasma PK parameters of DTG: Time of occurrence of Cmax (tmax) | 72 hours
Plasma PK parameters of DTG: Maximum observed concentration (Cmax) | 72 hours
Plasma PK parameters of DTG: Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration (AUC(0-t)) | 72 hours
Plasma PK parameters of DTG: Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC(0-infinity)) | 72 hours
Plasma PK parameters of DTG: Percentage of AUC(0-infinity) obtained by extrapolation (%AUCex) | 72 hours
Plasma PK parameters of DTG: Terminal phase half-life (t1/2) | 72 hours
Plasma PK parameters of DTG: Apparent clearance (CL/F) | 72 hours
Plasma PK parameters of DTG: Apparent terminal phase volume of distribution (Vz/F) | 72 hours

SECONDARY OUTCOMES:
Unbound concentration and unbound fraction in plasma of DTG at 3 hours post dose | 3 hours
Unbound concentration and unbound fraction in plasma of DTG at 24 hours post dose | 24 hours
Plasma ether glucuronide conjugate concentration | 72 hours
Grade 2 or higher adverse events | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Weller S, Borland J, Chen S, Johnson M, Savina P, Wynne B, Wajima T, Peppercorn AF, Piscitelli SC. Pharmacokinetics of dolutegravir in HIV-seronegative subjects with severe renal impairment. Eur J Clin Pharmacol. 2014 Jan;70(1):29-35. doi: 10.1007/s00228-013-1590-9. Epub 2013 Oct 6. PMID 24096683